CLINICAL TRIAL: NCT04353479
Title: Combined PD1 Inhibitor and Decitabine in Elderly Patients With Relapse and Refractory Acute Myeloid Leukemia : An Open-Label, Single-Arm, Phase 2 Study.
Brief Title: Combined PD1 Inhibitor and Decitabine in Elderly Patients With Relapse and Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Junmin Li, Director of Department of Hematology, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-AML-II-001
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: PD1 inhibitor; DNA methyltransferase inhibitor; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — camrelizumab; Immune Checkpoint Inhibitors; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab(SHR-1210) Combined With Decitabine (Experimental): Patients will be administered Camrelizumab(SHR-1210) at D1 and D15 and decitabine at D1-5. Treatment repeats every 28 days until disease progression or unacceptable toxicity.
  Interventions: Drug: Camrelizumab(SHR-1210); Drug: Decitabine

INTERVENTIONS:
Drug: Camrelizumab(SHR-1210) — A humanized monoclonal immunoglobulin
  Other Names: PD1 inhibitor
Drug: Decitabine — A DNA methyltransferase inhibitor
  Other Names: 5-aza-2- deoxycytidine

SUMMARY:
This is an open-label, single arm, phase 2 study to evaluate efficacy and safety of PD1 inhibitor Camrelizumab(SHR-1210) combined with DNA methyltransferase inhibitor decitabine in elderly patients with relapse and refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, 29 relapsed or refractory acute myeloid leukemia patients will be enrolled. Patients will be administered Camrelizumab(SHR-1210) at D1 and D15 and decitabine at D1-5. Treatment repeats every 28 days until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-75
* Relapsed and refractory patients with acute myeloid leukemia via morphology and immunology
* ECOG：0-2
* Life expectancy ≥ 3 months
* Adequate laboratory parameters during the screening period as evidenced by the following:

  1. Creatinine clearance≥30 mL/min and serum Creatinine ≤ 160µmol/L
  2. ALT and AST ≤ 3 × upper limit of normal (ULN)
  3. FEV1,FVC,DLCO ≥ 50% predicted value
  4. Left ventricular ejection fraction (LVEF) ≥ 40%, no symptomatic arrhythmia
  5. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

* Treatment-related AML
* Allergic to Camrelizumab, Decitabine, other monoclonal antibody or pharmaceutical excipients
* Use of immunosuppressive drug within 2 weeks before entering the group
* Abnormal liver and kidney function(does not meet the inclusion criteria)
* Suffering from heart failure
* Active tuberculosis or HIV positive
* Active hepatitis: Hepatitis B(HBsAg positive and HBV DNA≥500IU/mL), and hepatitis C(HCV RNA positive, abnormal liver function) ,Hepatitis B and hepatitis C infection in common.
* Active, known or suspected autoimmune disease. Subjects who were in a stable state without systemic immunosuppressive therapy were admitted
* Concurrent medical condition requiring the long-term use of immunosuppressive medications, or immunosuppressive doses of systemic corticosteroids > 10 mg/day topical prednisone or equivalent
* Suffer from other hematological neoplasm
* Known history of use other immune checkpoint inhibitor
* Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  CR, CRi, and morphologic leukemia-free state (MLFS)
Complete remission (CR) rate | 6 months
  Blast and promyelocytic leukemia less than 5% in bone marrow

SECONDARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  PFS is defined from the date of entry on study until disease progression, including treatment failure, relapse from CR, or death from any causes.
Overall survival (OS) | 2 years
  OS is defined for patients entering the study as time to death of all causes.
6-month overall survival rate | 6 months
  To evaluate overall survival rate at 6 months from study entry.
12-month overall survival rate | 12 months
  To evaluate overall survival rate at 12 months from study entry.
Hematological and non-hematological toxicity | 2 years
  Assessed according to the Common Terminology Criteria for Adverse Events Version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Li, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No